CLINICAL TRIAL: NCT03399682
Title: Incidence of Post Cystography Urinary Tract Infections in the Pediatric Population
Acronym: IUCPED
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Collaborators: CH Lisieux (Unknown); CH Avranches (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2017-A02445-48
Record Dates: First submitted 2018-01-08; First posted 2018-01-16 (Actual); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Urinary Infection
Keywords: cystography; pediatry; urinary infection
MeSH Terms: conditions — Urinary Tract Infections | interventions — Cystography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Incidence of Post Cystography Urinary Tract Infections: all children less than 16 years having cystography
  Interventions: Diagnostic Test: cystography

INTERVENTIONS:
Diagnostic Test: cystography — observationnal study

SUMMARY:
Cystography is a frequent pediatric examination, although indications have been recently restricted .

Current indications in our center are:

* The occurrence of 2 episodes of acute pyelonephritis
* or 1 episode of pyelonephritis if dilatation of the pelvic ureter> 5 mm for male children Urinary tract infections that occurred in the month following this test are considered secondary to cystography.

However, no recent study has investigated the prevalence of urinary tract infections post cystography.

There is no recent epidemiological data on this risk of infection, especially since the management of infections has changed and aseptic precautions during retrograde cystography have evolved with most of the time coverage. antibiotic.

The main objective of this multi-center epidemiological prospective study is to perform a recent analysis of the retrograde post-cystographic urinary tract infection rate.

Material and methods:

Epidemiological, observational, multicenter, prospective study over a period from January 2018 to January 2019. No therapeutic modification will be undertaken at the end of the study.

Parents will be called one months after the exam to check if their child had a urinary infection.

DETAILED DESCRIPTION:
Cystography is a frequent examination, performed in the context of acute pyelonephritis.

However, its realization has decreased significantly, in particular because of the invasive aspect and urinary infections identified retrospectively. (1) (2) (3) (4)

The only indications to the University Hospital of Caen are:

* 2 acute pyelonephritis
* or 1 acute pyelonephritis if the pelvic ureter> 5 mm in boys

There are 2 techniques for performing cystography:

* The first is retrograde cystography which is performed most often in our center, and whose disadvantages are the traumatic effect and the increased risk of urinary tract infection. (5)
* The 2nd technique is cystography by the pubic route for which the bladder must be full, which is difficult in newborns not clean The advantages, however, are the ability to take urine directly into the bladder for bacteriological and cytological analysis, to be less traumatic and totally sterile. (5) (6)

Urinary tract infections during the month following cystography are considered secondary to cystography. (7) They are estimated at 6% in old studies (7) However, there is no recent study on the prevalence of urinary tract infections after cystography (article (7): 6%: Complications of voiding cystourethrography in the evaluation of infants with prenatally detected hydronephrosis, The Journal of Urology, 162, 1221-1223, september 1999)

The main objective of our study is therefore to have recent data on the rate of retrograde post cystographic urinary tract infections in the month following the examination.

The secondary objectives are to analyze the rate of urinary tract infections according to age, sex, indications, and circumstances.

Material and method:

Epidemiological, observational, multicenter, prospective study over a period from January 2018 to January 2019. No therapeutic modification will be undertaken at the end of the study.

Included patients are all children under 16 years of age with retrograde cystography and excluded patients are children over 16 years old and those with ongoing infection.

During the realization of the cystography the information required for the study will be noted, namely:

* name
* age
* sex
* indication of cystography / ultrasound data
* antibiotic preventive or not
* results of cystography
* antibiotic post cystography or not
* parental consent and parents' contact information

Clear, fair, and appropriate information about the study is then given to the parents.

They are informed, that with their authorization, they will receive a call to a month of the cystography to know if their child presented a urinary infection (fever, BU and ECBU positive) after the gestexamure.

Their written consent is collected. The data collected after the telephone passages are listed in a table and will be analyzed at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* age: less than 16 years
* had a retrograd cystography

Exclusion Criteria:

* older than 16 years
* urinary infection in progress

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: all patients under the age of 16 who have had retrograde cystograph
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-01-03 (Actual); Primary Completion 2018-02-03 (Estimated); Study Completion 2019-01-31 (Estimated)

PRIMARY OUTCOMES:
recent analysis of urinary post cystography infection rate in the pediatric population | 1 month
  fievre, urine test strip, CBEU

SECONDARY OUTCOMES:
infection rate epidemiology | 1 month
  age, sexe; indication of the test

CONTACTS AND LOCATIONS:
Overall Officials: Kassel christophe, Principal Investigator — CHU CAEN
Locations (1):
- Caen University Hospital, Caen, France

IPD SHARING:
Plan to Share IPD: No